CLINICAL TRIAL: NCT01160835
Title: Comparison of Quadriceps-sparing Minimally Invasive and Medial Parapatellar Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ching-Chuan Jiang, Professor, Department of Orthopaedic Surgery of National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9561705022
Record Dates: First submitted 2010-07-01; First posted 2010-07-12 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-06

CONDITIONS: Osteoarthritis
Keywords: total knee arthroplasty; minimally invasive; quadriceps-sparing; Quadriceps-sparing total knee arthroplasty
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadriceps-sparing total knee arthroplasty (Experimental): Quadriceps-sparing arthrotomy with side-cutting instruments
  Interventions: Procedure: total knee arthroplastyinstruments
- Medial parapatellar total knee arthroplasty (Active Comparator): Medial parapatellar arthrotomy with front-cutting instruments
  Interventions: Procedure: total knee arthroplastyinstruments

INTERVENTIONS:
Procedure: total knee arthroplastyinstruments — Quadriceps-sparing arthrotomy with side-cutting instruments

SUMMARY:
Quadriceps-sparing minimally invasive total knee arthroplasty (TKA) with side-cutting instruments has been proposed to limit surgical dissection without compromising the surgical outcome. We conducted a prospective, randomized study to compare the outcomes of quadriceps-sparing TKA with conventional medial parapatellar TKA, with two-year follow-up.

We hypothesize that the quadriceps-sparing arthrotomy would not outperform the conventional medial parapatellar arthrotomy in TKA, in terms of postoperative recovery of quadriceps muscle strength, alignment of the prosthetic knee, and clinical outcome.

DETAILED DESCRIPTION:
Eighty primary TKAs in sixty patients of osteoarthritis constituted this study. Patients were randomly assigned to either quadriceps-sparing (QS, 40 knees) or medial parapatellar (MP, 40 knees) group. All surgeries were designed to set the prosthesis with thefemoral component alignment of 7º valgus and the tibial component alignment perpendicular to tibial shaft. Outcome variables included knee function defined by Hospital for Special Surgery knee score, quadriceps muscle strength measured by isokinetic dynamometer, pain indicated on visual analogue scale, range of motion, and post-operative alignment measured on plain radiograph.

ELIGIBILITY:
Inclusion Criteria:

* advanced osteoarthritis with radiograph-evident narrowing of joint gap,
* with persistent symptoms after conservative treatment for at least 6 months, and
* patients' intention to receive the prosthetic TKA.

Exclusion Criteria:

* the knees with excessive deformity of femorotibial angle exceeding 15° varus or 10° valgus,
* flexion contracture exceeding 15°,
* active infection involving the knees, or
* knees received previous surgery.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-05; Primary Completion 2006-02 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To compare the clinic and functional outcomes of total knee arthroplasty (TKA) respectively through a quadriceps-sparing (QS) approach and a MIS medial parapatellar (MP) approach | 2 years
  Perioperative parameters: operative time, blood loss, Doses of narcotics for pain control, peri-operative complications Postoperative parameters: VAS, range of motion, knee functional score, isokinetic studies, radiographic alignment, complications

SECONDARY OUTCOMES:
To compare the survival and functional outcomes of total knee arthroplasty (TKA) respectively through a quadriceps-sparing (QS) approach and a MIS medial parapatellar (MP) approach at 2-year follow-up. | 5 and 10 years
  Postoperative parameters: VAS, range of motion, knee functional score, isokinetic studies, radiographic alignment and failure rate of knee prothesis

CONTACTS AND LOCATIONS:
Overall Officials: Hongsen Chiang, M.D., Ph.D, Principal Investigator — Department of orthopedic surgery of National Taiwan University Hospital
Locations (1):
- Department of Orthopedic Surgery, National Taiwan University Hospital, Taipei, Taiwan